CLINICAL TRIAL: NCT05800223
Title: Prospective, Multicenter, Randomized Controlled, Phase III Clinical Study of Armatinib Alone or in Combination With Stereotactic Body Radiotherapy (SRT) for First-line Treatment of Brain Metastases From EGFR-mutated Non-small Cell Lung Cancer
Brief Title: Armatinib Alone or in Combination With SRT for Brain Metastases EGFR-mutated Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Cancer Hospital, China (Other)
Responsible Party: Principal Investigator, Fan Min, Clinical Professor, Shanghai Cancer Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUSCC-20230323
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Non-small Cell Lung Cancer Metastatic
MeSH Terms: interventions — aumolertinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GroupA (Experimental): Intracranial stereotactic radiotherapy (27-40 Gy/3-5f) was administered to all intracranial lesions on the first day of oral administration of Almonertinib
  Interventions: Drug: Almonertinib; Radiation: SBRT
- GroupB (Experimental): Two successive MR enhancements after oral administration of Almonertinib suggest that intracranial lesions are maximally remission, and stereotactic body radiotherapy is given to all lesions (27-40Gy/3-5f)
  Interventions: Drug: Almonertinib; Radiation: SBRT
- GroupC (Experimental): oral administration of Almonertinib
  Interventions: Drug: Almonertinib

INTERVENTIONS:
Drug: Almonertinib — The dosage is 110 mg/day (2 tablets/day) orally once a day
Radiation: SBRT — SRT, 27Gy-40Gy/3-5f
  Arms: GroupA; GroupB

SUMMARY:
Objective:Patients with asymptomatic or minimally symptomatic Stage IV EGFR-positive NSCLC with baseline intracranial metastases.

Aim: To investigate the timing, efficacy and safety of radiotherapy in patients with EGFR positive brain metastases treated with armatinib alone or combined with stereotactic radiotherapy.

Method: Almonertinib: specification 55mg/tablet; The dosage is 110 mg / day (2 tablets / day) orally once a day; SBRT: 3-5 doses of 27-40 Gy

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 years or older (including 18 years) and up to 75 years (including 75 years)
2. histologically confirmed NSCLC (by AJCC 8th edition lung cancer staging criteria)
3. asymptomatic or minimally symptomatic brain metastases (i.e., headache, nausea, or seizures responding to dexamethasone/analgesic/antiepileptic agents at a stable drug dose for at least 3 days);
4. brain metastases must meet the following criteria on diagnostic MRI: at least one lesion that can be classified as measurable disease according to RANO-BM, ≤ 10 brain or brainstem metastases
5. epidermal growth factor receptor (EGFR) exon 19 deletion or exon 21 (L858R) substitution mutation (alone or in combination with other EGFR mutations);
6. no prior systemic therapy other than neoadjuvant therapy, adjuvant therapy, or concurrent chemotherapy for more than 3 months prior to study entry
7. Eastern Cooperative Oncology Organization Group (ECOG) physical status score of 0 or 1 and no worsening in the previous 2 weeks, with a minimum expected survival of 12 weeks.
8. good hematopoietic function, defined as absolute neutrophil count ≥ 1.5 × 109 /L, platelet count ≥ 100 × 109 /L, and hemoglobin ≥ 90 g/L [no transfusion or erythropoietin (EPO-dependent) within 7 days
9. good coagulation, defined as an international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN; if the subject is on anticoagulation therapy, as long as the PT is within the proposed range of anticoagulant medication
10. good liver function, defined as a total bilirubin level ≤ 1.5 times the upper limit of normal (ULN); glutathione transaminase (AST) and glutamate transaminase (ALT) levels ≤ 2.5 times the ULN for patients without liver metastases; and AST and ALT levels ≤ 5 times the ULN for patients with documented liver metastases
11. good renal function, defined as serum creatinine ≤ 1.5 times ULN or calculated creatinine clearance ≥ 60 ml/min; urine protein less than 2+ on routine urine examination, or 24-hour urine protein quantification < 1 g
12. Women of childbearing potential should have a negative urine or serum pregnancy test within 3 days prior to receiving the first dose of study drug (Week 1, Day 1).
13. male patients should be using barrier contraception (i.e., condoms) from screening until 6 months after discontinuation of study treatment
14. Subjects will voluntarily participate and sign an informed consent in writing.

Exclusion Criteria:

1. Received any of the following treatments:

   1. Currently participating in an interventional clinical study treatment or received another study drug within 4 weeks prior to the first dose
   2. Received palliative intracranial radiation therapy prior to the first dose
   3. Patient has undergone major surgery (including biopsy) or major trauma within 4 weeks prior to the first dose of study drug; patients who are expected to require major surgery during the study period
   4. Patients previously treated with EGFR-TKI.
2. patients with NSCLC EGFR driver gene negative or known severe allergic reactions (≥ grade 3) to TKIs drugs;
3. patients who are unable to undergo MR examination
4. brain metastases requiring surgical decompression;
5. the presence of a previous solid organ or hematologic transplant; clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction; the presence of clinically uncontrollable pleural effusion/peritoneal effusion
6. malignancy other than non-small cell lung cancer within 5 years prior to enrollment, excluding adequately treated carcinoma in situ of the cervix, basal cell or squamous epithelial cell skin cancer of the skin, localized prostate cancer after radical surgery, and ductal carcinoma in situ of the breast;
7. having unremitting residual toxicity of prior therapy greater than CTCAE grade 1 at the time of initiation of study treatment, with the exception of alopecia and grade 2 neurotoxicity from prior chemotherapy;
8. have any serious or poorly controlled systemic disease, such as active bleeding-prone body or active infection, as judged by the investigator. Chronic illnesses that do not require exclusion;
9. the known presence of a psychiatric illness or substance abuse condition that may have an impact on compliance with trial requirements
10. any serious or uncontrolled ocular pathology that, in the judgment of the physician, may increase the safety risk to the patient
11. a known history of human immunodeficiency virus (HIV) infection (i.e., HIV 1/2 antibody positive)
12. patients who, in the judgment of the investigator, are likely to be poorly compliant with the procedures and requirements of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
iPFS | up to 12 months
  Intracranial to time to disease progression

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No